CLINICAL TRIAL: NCT02732340
Title: Triple-branch Stent Graft Placement for the Treatment of Acute DeBakey I Aortic Dissection: A Prospective, Single-center, Open-label, Non-controlled Clinical Trial
Brief Title: Triple-branch Stent Graft Placement for the Treatment of Acute DeBakey I Aortic Dissection
Acronym: TBSGPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, The director of the department of cardiovascular surgery, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLW2015AD
Record Dates: First submitted 2015-11-15; First posted 2016-04-08 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Acute Aortic Dissection
Keywords: triple-branched stent graft; the occluded rate of false lumen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- triple-branched stent graft (Experimental): The triple-branched stent graft was a branched 1-piece graft and included a main stent graft and 3 sidearm stent grafts (Yuhengjia Science and Technology, Corp, Ltd, Beijing, China). The main stent graft and sidearm stent grafts were individually mounted on 4 catheters and restrained by 4 silk sutures .The triple-branched stent graft was inserted into the true lumens of the aortic arch and proximal descending aorta; the three vascular stent branches were then grafted into the corresponding true lumens of the aortic arch branch vessels followed by the sequential release of the vascular stent backbone and the branch stents in the left subclavian artery, the left common carotid artery, and the innominate artery.
  Interventions: Procedure: triple-branched stent graft

INTERVENTIONS:
Procedure: triple-branched stent graft — place the triple-branched stent graft into the aortic arch, descending aorta ,the left subclavian artery, the left common carotid artery, and the innominate artery.

SUMMARY:
The purpose of this study is to evaluate triple-branched stent placement in the treatment of acute DeBakey I aortic dissection . The investigators design a prospective, single-center, open-label, non-controlled clinical trial.

DETAILED DESCRIPTION:
From November 2015, 150 consecutive patients with acute DeBakey I aortic dissection were treated with triple-branched stent placement.

In all cases, surgery was performed under general anesthesia with tracheal intubation and cardiopulmonary bypass (CPB). During surgery arterial pressures at the upper and lower limbs were monitored. An esophageal echocardiography probe was placed routinely, and a sternal incision was performed. To establish CPB, the perfusion tube was placed in the right axillary artery and the drainage tube was placed in the superior and inferior vena cava through the right atrium. The CPB flow rate was of 2.4-2.6 L/kg/min. Intermittent cold blood cardioplegia was perfused through the left and right coronary arteries for myocardial protection.

The innominate artery and the left common carotid artery were fully isolated during the CPB cooling process. The ascending aorta proximal to the innominate artery was occluded, and the ascending aorta was transected slightly above the sinus tube connection; the left and right coronary arteries were directly perfused with blood-containing cold cardioplegia. Proximal procedures such as aortic valve repair, sinus reconstruction, and root replacement were performed first. Afterwards, the stumps were reconstructed. The reconstructed aortic root stump was anastomosed with a Dacron graft of corresponding size using 4-0 polypropylene suture (ascending aorta replacement). The nasopharyngeal temperature was then decreased to 25° (usually a rectal temperature of 27-29°C), the aortic perfusion flow was set to 10-15 ml/kg/min, and the innominate artery and the left common carotid artery were occluded 5-6 cm above the aortic arch. The aortic occlusion clamp was removed and a half aortic arch transection was made about 2 cm proximal to the innominate artery. Through the incision, the true lumens of the aortic arch, the proximal descending aorta, and the three aortic branches were identified. The triple-branched stent graft was inserted into the true lumens of the aortic arch and proximal descending aorta; the three stent graft branches were then placed into the corresponding true lumens of the aortic arch branch vessels followed by the sequential release of the vascular stent backbone and the branch stents in the left subclavian artery, the left common carotid artery, and the innominate artery. A catheter with a balloon or a probe was used to expand the vascular stents and the graft and branches were examined for kinks or folding of the backbone. A sandwich reconstruction was performed between the aortic stump, the aortic external Dacron graft, and the proximal stentless suture zone of the intraluminal artificial vessel backbone. The reconstructed stump was anastomosed with the Dacron graft that replaced the ascending aorta using 4-0 polypropylene suture. The occlusions of the left common carotid artery and the innominate artery were then relieved, and air was fully flushed out from the heart and the aorta. The right axillary artery perfusion was stopped, and systemic perfusion via an aortic perfusion tube at the artificial portion of the ascending aorta was performed. The patient was rewarmed after oxygen debt repayment, followed by the cardiac resuscitation.

Telephone contact was maintained with the patients after discharge. At 3,6,12 months postoperatively , patients received a follow-up examination, chest radiography, echocardiography, bilateral carotid artery Doppler examinations and CT angiography (CTA) examinations Numerical data were expressed as percentages. Quantitative data were expressed as mean ± standard deviation. The primary end point is the occluded rate of the false lumen one year postoperatively. The secondary end point are the survive rate ,complication, reoperation rate, the growth rate of thoracic descending aorta, security index perioperatively, life quality postoperatively.Statistical analysis were performed with SPSS 11.5 software. A value of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age<65 years;
* acute DeBakey I aortic dissection is confirmed by CTA; cardiac function is NYHA(New York Heart Association) I-II;
* the onset time< 2 weeks;
* the patient or family members can understand the research plan and will participate in this study and provide a written informed consent

Exclusion Criteria:

* Dissection involved the superior mesenteric artery, renal artery and coronary artery, which affect the body's viscera function seriously. The principal researcher from different centre need judge the patients' condition.
* there is a serious complication of nervous system, such as coma, paraplegia, etc
* pregnant or lactating women
* anyone with severe emphysema, interstitial pneumonia or ischemic heart disease cannot tolerate surgery
* subjects with contraindications of heart surgery, anesthesia and extracorporeal circulation
* subjects had significant or progressive of heart disease, according to the experience of the researchers,whose life expectancy is less than 1 year, or placement of triple- branched stent graft will induce unacceptable risk to the subjects;
* anyone with serious mental illness, drug abuse, alcoholism, prison inmates, a lack of ability to care for, or can not express the informed consent
* subjects are incompliance or can't complete the research
* anyone is involved in the other clinical trial
* other reasons are not suitable for clinical trials, according to the researchers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
the occluded rate of false lumen by CTA | one year postoperatively

SECONDARY OUTCOMES:
the survive rate by the questionaire | 3 months, 6 months, 12 months postoperatively
complication by the case report | 1 months postoperatively
reoperation rate by the case report | 1 year postoperatively
the growth rate of thoracic descending aorta by CTA | 3 months, 6 months, 12 months postoperatively
life quality by the questionaire | 3 months, 6 months, 12 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- the Department of Cardiovascular Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Estrera AL, Miller CC 3rd, Huynh TT, Porat E, Safi HJ. Neurologic outcome after thoracic and thoracoabdominal aortic aneurysm repair. Ann Thorac Surg. 2001 Oct;72(4):1225-30; discussion 1230-1. doi: 10.1016/s0003-4975(01)02971-x. PMID 11603441
- [Background] Chiappini B, Schepens M, Tan E, Dell' Amore A, Morshuis W, Dossche K, Bergonzini M, Camurri N, Reggiani LB, Marinelli G, Di Bartolomeo R. Early and late outcomes of acute type A aortic dissection: analysis of risk factors in 487 consecutive patients. Eur Heart J. 2005 Jan;26(2):180-6. doi: 10.1093/eurheartj/ehi024. Epub 2004 Dec 7. PMID 15618075
- [Background] Trimarchi S, Nienaber CA, Rampoldi V, Myrmel T, Suzuki T, Mehta RH, Bossone E, Cooper JV, Smith DE, Menicanti L, Frigiola A, Oh JK, Deeb MG, Isselbacher EM, Eagle KA; International Registry of Acute Aortic Dissection Investigators. Contemporary results of surgery in acute type A aortic dissection: The International Registry of Acute Aortic Dissection experience. J Thorac Cardiovasc Surg. 2005 Jan;129(1):112-22. doi: 10.1016/j.jtcvs.2004.09.005. PMID 15632832
- [Background] Rampoldi V, Trimarchi S, Eagle KA, Nienaber CA, Oh JK, Bossone E, Myrmel T, Sangiorgi GM, De Vincentiis C, Cooper JV, Fang J, Smith D, Tsai T, Raghupathy A, Fattori R, Sechtem U, Deeb MG, Sundt TM 3rd, Isselbacher EM; International Registry of Acute Aortic Dissection (IRAD) Investigators. Simple risk models to predict surgical mortality in acute type A aortic dissection: the International Registry of Acute Aortic Dissection score. Ann Thorac Surg. 2007 Jan;83(1):55-61. doi: 10.1016/j.athoracsur.2006.08.007. PMID 17184630
- [Background] Crawford ES, Kirklin JW, Naftel DC, Svensson LG, Coselli JS, Safi HJ. Surgery for acute dissection of ascending aorta. Should the arch be included? J Thorac Cardiovasc Surg. 1992 Jul;104(1):46-59. PMID 1614214
- [Background] Ohtsubo S, Itoh T, Takarabe K, Rikitake K, Furukawa K, Suda H, Okazaki Y. Surgical results of hemiarch replacement for acute type A dissection. Ann Thorac Surg. 2002 Nov;74(5):S1853-6; discussion S1857-63. doi: 10.1016/s0003-4975(02)04133-4. PMID 12440680
- [Background] Hirotani T, Nakamichi T, Munakata M, Takeuchi S. Routine extended graft replacement for an acute type A aortic dissection and the patency of the residual false channel. Ann Thorac Surg. 2003 Dec;76(6):1957-61. doi: 10.1016/s0003-4975(03)01325-0. PMID 14667621
- [Background] Takahara Y, Sudo Y, Mogi K, Nakayama M, Sakurai M. Total aortic arch grafting for acute type A dissection: analysis of residual false lumen. Ann Thorac Surg. 2002 Feb;73(2):450-4. doi: 10.1016/s0003-4975(01)03422-1. PMID 11845858
- [Background] Urbanski PP, Siebel A, Zacher M, Hacker RW. Is extended aortic replacement in acute type A dissection justifiable? Ann Thorac Surg. 2003 Feb;75(2):525-9. doi: 10.1016/s0003-4975(02)04378-3. PMID 12607666
- [Background] Khan IA, Nair CK. Clinical, diagnostic, and management perspectives of aortic dissection. Chest. 2002 Jul;122(1):311-28. doi: 10.1378/chest.122.1.311. PMID 12114376
- [Background] Pochettino A, Brinkman WT, Moeller P, Szeto WY, Moser W, Cornelius K, Bowen FW, Woo YJ, Bavaria JE. Antegrade thoracic stent grafting during repair of acute DeBakey I dissection prevents development of thoracoabdominal aortic aneurysms. Ann Thorac Surg. 2009 Aug;88(2):482-9; discussion 489-90. doi: 10.1016/j.athoracsur.2009.04.046. PMID 19632398
- [Background] Kim JB, Chung CH, Moon DH, Ha GJ, Lee TY, Jung SH, Choo SJ, Lee JW. Total arch repair versus hemiarch repair in the management of acute DeBakey type I aortic dissection. Eur J Cardiothorac Surg. 2011 Oct;40(4):881-7. doi: 10.1016/j.ejcts.2010.12.035. Epub 2011 Feb 18. PMID 21315615
- [Background] Zierer A, Voeller RK, Hill KE, Kouchoukos NT, Damiano RJ Jr, Moon MR. Aortic enlargement and late reoperation after repair of acute type A aortic dissection. Ann Thorac Surg. 2007 Aug;84(2):479-86; discussion 486-7. doi: 10.1016/j.athoracsur.2007.03.084. PMID 17643619
- [Background] Halstead JC, Meier M, Etz C, Spielvogel D, Bodian C, Wurm M, Shahani R, Griepp RB. The fate of the distal aorta after repair of acute type A aortic dissection. J Thorac Cardiovasc Surg. 2007 Jan;133(1):127-35. doi: 10.1016/j.jtcvs.2006.07.043. Epub 2006 Dec 4. PMID 17198797
- [Background] Park KH, Lim C, Choi JH, Chung E, Choi SI, Chun EJ, Sung K. Midterm change of descending aortic false lumen after repair of acute type I dissection. Ann Thorac Surg. 2009 Jan;87(1):103-8. doi: 10.1016/j.athoracsur.2008.09.032. PMID 19101279
- [Background] Jakob H, Tsagakis K, Tossios P, Massoudy P, Thielmann M, Buck T, Eggebrecht H, Kamler M. Combining classic surgery with descending stent grafting for acute DeBakey type I dissection. Ann Thorac Surg. 2008 Jul;86(1):95-101. doi: 10.1016/j.athoracsur.2008.03.037. PMID 18573404
- [Background] Uchida N, Shibamura H, Katayama A, Shimada N, Sutoh M, Ishihara H. Operative strategy for acute type a aortic dissection: ascending aortic or hemiarch versus total arch replacement with frozen elephant trunk. Ann Thorac Surg. 2009 Mar;87(3):773-7. doi: 10.1016/j.athoracsur.2008.11.061. PMID 19231387
- [Background] Gorlitzer M, Weiss G, Meinhart J, Waldenberger F, Thalmann M, Folkmann S, Moidl R, Grabenwoeger M. Fate of the false lumen after combined surgical and endovascular repair treating Stanford type A aortic dissections. Ann Thorac Surg. 2010 Mar;89(3):794-9. doi: 10.1016/j.athoracsur.2009.11.054. PMID 20172130
- [Result] Chen LW, Dai XF, Lu L, Zhang GC, Cao H. Extensive primary repair of the thoracic aorta in acute type a aortic dissection by means of ascending aorta replacement combined with open placement of triple-branched stent graft: early results. Circulation. 2010 Oct 5;122(14):1373-8. doi: 10.1161/CIRCULATIONAHA.110.946012. Epub 2010 Sep 20. PMID 20855660
- [Result] Chen LW, Wu XJ, Lu L, Zhang GC, Yang GF, Yang ZW, Dong Y, Cao H, Chen Q. Total arch repair for acute type A aortic dissection with 2 modified techniques: open single-branched stent graft placement and reinforcement of the dissected arch vessel stump with stent graft. Circulation. 2011 Jun 7;123(22):2536-41. doi: 10.1161/CIRCULATIONAHA.110.008656. Epub 2011 May 16. PMID 21576657